CLINICAL TRIAL: NCT07165899
Title: Effects of Exposure to a Single-electrode Electroencephalography-guided Binaural Beat Audio Track on Sustained Attention and Subjective Well-being Among Healthy Adults: a Randomized, Double-blinded, Sham-controlled Repeated-measures Crossover Trial
Brief Title: Effects of Exposure to a Single-electrode Electroencephalography-guided Binaural Beat Audio Track on Sustained Attention and Subjective Well-being Among Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Principal Investigator, Samudani Dhanasekara, Assistant Professor, Texas Tech University Health Sciences Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB-FY2024-286
Record Dates: First submitted 2025-08-14; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Psychomotor Speed; Sustained Attention; Inhibitory Control; Memory Encoding; Well-being

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, sham-controlled, repeated-measures crossover design
Who Masked: Participant, Investigator
Masking Description: Both participants and research staff will be blinded to condition; randomization and condition assignment are automated within the PsychoPy script.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EEG-Guided Binaural Beat Audio (Experimental): 30-minute audio session with dynamic frequency adjustments based on real-time EEG feedback
  Interventions: Behavioral: EEG-Guided Binaural Beat Audio
- Sham Control (Sham Comparator): 30-minute audio session with identical tones presented to both ears, EEG monitored but not used for frequency adjustment
  Interventions: Behavioral: Sham Control

INTERVENTIONS:
Behavioral: EEG-Guided Binaural Beat Audio — 30-minute audio session with dynamic frequency adjustments based on real-time EEG feedback
  Arms: EEG-Guided Binaural Beat Audio
Behavioral: Sham Control — 30-minute audio session with identical tones presented to both ears (no binaural beat), EEG monitored but not used for frequency adjustment
  Arms: Sham Control

SUMMARY:
This study aims to explore the potential of binaural beats, adjusted in real-time via EEG feedback, to positively influence brain states related to relaxation, focus, and cognitive performance. The investigators are examining how these auditory techniques can improve memory, attention, and overall subjective well-being.

DETAILED DESCRIPTION:
With the existence of a strong evidence base regarding audio-assisted relaxation, audio products are widely used globally to achieve relaxed and focused mental states. The utility of audio for achieving relaxed mental states has revolutionized with the advent of the concept of binaural beats, an auditory phenomenon that is induced by separately presenting two tones of different frequencies to each ear. The superior olivary nucleus of the midbrain computes the difference between the two tones, and with time, the brain state is expected to synchronize with the difference in the frequencies presented to the two ears. Binaural beats are widely used to achieve relaxed mental states for applications including improved memory, enhanced relaxation, augmented hypnotherapy, improved sleep quality, creating and breaking habits, addiction therapy, and enhanced cognitive performance with limited empirical support.

Electroencephalography (EEG) is a well-established technique for recording the electrical activity of the brain. This is conventionally achieved through the placement of multiple electrodes across the scalp, allowing for the detection of the brain's spontaneous electrical activity over a period of time. EEG measures voltage fluctuations resulting from ionic current flows within the neurons of the brain. Single-electrode electroencephalography simplifies the conventional approach by using one electrode placed at a strategic location on the scalp. When recorded over the pre-frontal cortex, this method allows for capturing the electrical activity of the brain's frontal lobe, which is responsible for high-level cognitive functions and behavior. EEG waves are typically divided into bandwidths known as frequency bands. These are characterized based on their frequency, which is measured in cycles per second (Hz), and include:

Delta waves (0 to 4 Hz): Associated with deep sleep and certain pathological conditions.

Theta waves (4.1 to 8 Hz): Linked to drowsiness, early stages of sleep, and meditation.

Low Alpha waves (8.1 to 10 Hz): Related to relaxed, calm, and resting states. High Alpha waves (10.1 to 14 Hz): Often associated with a state of wakeful relaxation.

Low beta waves (14.1-20 Hz): Associated with arousal, active thought, concentration, complex thought High beta waves (20.1-32 Hz): Associated with heightened arousal, hyperactive thought, hypervigilance, and states of anxiety/panic While the brain produces all of these wave types simultaneously, typically, one frequency band is dominant at any given time, reflecting the predominant brain state. For instance, during deep sleep, delta waves predominate, while during active concentration, beta waves are more prominent.

The Frequency-Following Response (FFR) is a neurophysiological mechanism where brain EEG activity synchronizes with auditory frequency stimuli. This synchronization is particularly evident with binaural beats. While many studies have supported the notion that binaural beats, via FFR, can induce desired brain states that are particularly for relaxation (e.g., increased high alpha activity), increased receptivity for hypnotic suggestions (e.g., heightened low alpha or theta activity), as well as induce sleep and improve the quality of sleep. However, other studies have challenged this notion, supported by not observing a significant FFR when the brains were stimulated for a duration of < 5 minutes with one binaural beat frequency falling within a particular band at a given time. In fact, delivering binaural beats to participants, regardless of their current brain state, could result in discomfort, headaches, and dizziness.

The proposed study aims to overcome this limited efficacy of a static binaural beat frequency in eliciting an FFR by guiding the delivered binaural beat frequency with real-time feedback obtained from a single-electrode EEG. Based on the current biological understanding of FFR, the investigators propose to conduct a randomized, double-blinded, sham-controlled repeated-measures crossover trial to answer the following research questions:

1. Can a dynamic binaural beat frequency implemented with single-electrode EEG guidance elicit an FFR to guide the predominant EEG frequency of an individual to a target low alpha state?
2. Can a target low-alpha state achieved with the EEG feedback be sustained while the binaural beats are delivered at the target low-alpha frequency?
3. Will guiding the brain to the low-alpha state and maintaining it for up to 15 minutes in the target low-alpha state be associated with improvements in

   1. subjective perception of relaxation, sleepiness, focus, performance on cognitive tasks, and overall well-being
   2. objectively measured speed of reacting to stimuli, attention, inhibitory control (i.e., decreased impulsivity), and better memory encoding in a stop-signal reaction task
   3. objective performance in a Go-No-Go task
   4. objective performance in a graded novelty encoding task

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults (age > 18 years)

Exclusion Criteria:

* Cognitive impairment (self-reported)
* Gross visual, auditory, or motor impairments; severe physical, psychiatric, or neurological impairments
* History of epilepsy, seizures, or seizure-like episodes
* History of intracranial lesions, stroke, traumatic brain injury, neoplasms, cranial surgery, or foreign bodies
* Current daily alcohol or substance abuse
* Current daily use of medications affecting EEG activity (e.g., anti-epileptics, opioids) or lowering seizure threshold
* Self-reported auditory hypersensitivity or prior adverse effects from audio stimulation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-08-16 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Stop Signal Reaction Time | Baseline (At visit 2 or 3, immediately prior to 30-minute intervention/control audio session) and immediately post-intervention/control audio session (within 10 minutes after completion of session).
  Estimated time (milliseconds) required to inhibit a prepotent response following a stop signal, derived from the integration method. Lower values indicate better inhibitory control.
Reaction Time on Novelty Encoding Task | Baseline (at visit 2 or 3, immediately prior to 30-minute intervention/control audio session) and immediately post-intervention/control audio session (within 20 minutes after completion of session).
  Mean response latency (seconds) during the novelty encoding task recognition phase. Lower values indicate faster information retrieval and decision speed without implying a speed-accuracy trade-off. The unit of measurement is in seconds.
Predominant Frequency and Frequency Band from a Single Prefrontal Electrode | The duration of the audio intervention was 30 minutes. Predominant frequency and frequency bands were measured as baseline, 5, 10, 15, 20, 25 minutes, and at the end of the session (at 30 minutes).
  EEG data were segmented into epochs and subjected to quality control procedures. For each epoch, sample entropy was calculated as a measure of signal irregularity. Epochs with entropy values above the 75th percentile were classified as high-noise and excluded from further analysis. The remaining epochs were standardized by z-scoring, transformed to the frequency domain, and then summarized into standard bands (delta: 0.5-4 Hz, theta: 4-8 Hz, low-alpha: 8-10 Hz, high-alpha: 10-12 Hz, low-beta: 12-18 Hz, high-beta: 18-32 Hz) to facilitate comparison across participants and conditions.

SECONDARY OUTCOMES:
Visual Analogue Scale - Subjective Relaxation | Baseline (At visit 2 or 3, immediately prior to 30-minute intervention/control audio session) and immediately post-intervention/control audio session (within 20 minutes after completion of session).
  Self-reported relaxation, rated on a visual analogue scale (0-100; higher scores indicate greater relaxation).
Visual Analogue Scale - Sleepiness | Baseline (At visit 2 or 3, immediately prior to 30-minute intervention/control audio session) and immediately post-intervention/control audio session (within 20 minutes after completion of session).
  100 mm VAS, anchored at 0 ("Fully awake") and 100 ("Extremely sleepy"). Higher scores = greater sleepiness.
Visual Analogue Scale - Focus | Baseline (At visit 2 or 3, immediately prior to 30-minute intervention/control audio session) and immediately post-intervention/control audio session (within 20 minutes after completion of session).
  100 mm VAS, anchored at 0 ("Not focused at all") and 100 ("Extremely focused"). Higher scores = greater perceived focus.
Visual Analogue Scale - Cognitive Performance | Baseline (At visit 2 or 3, immediately prior to 30-minute intervention/control audio session) and immediately post-intervention/control audio session (within 20 minutes after completion of session).
  100 mm VAS, anchored at 0 ("Very poor performance") and 100 ("Excellent performance"). Higher scores = better perceived cognitive performance.
Visual Analogue Scale - Overall Well-Being | Baseline (At visit 2 or 3, immediately prior to 30-minute intervention/control audio session) and immediately post-intervention/control audio session (within 20 minutes after completion of session).
  100 mm VAS, anchored at 0 ("Very poor well-being") and 100 ("Excellent well-being"). Higher scores = better well-being.
Hit Rate of Novelty Encoding Task | Baseline (At visit 2 or 3, immediately prior to 30-minute intervention/control audio session) and immediately post-intervention/control audio session (within 20 minutes after completion of session).
  Proportion of targets correctly identified as "seen." Range 0-1; higher values indicate better recognition sensitivity. The unit of measurement is in proportion (0-1).
False Alarm Rate of Novelty Encoding Task | Baseline (At visit 2 or 3, immediately prior to 30-minute intervention/control audio session) and immediately post-intervention/control audio session (within 20 minutes after completion of session).
  Proportion of non-targets incorrectly endorsed as "seen." Range 0-1; lower values indicate better discrimination (fewer false positives). The unit of measurement is in proportion (0-1).

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, TX, USA, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data may be shared with qualified researchers upon a reasonable request and after obtaining institutional approval.